CLINICAL TRIAL: NCT04954820
Title: A Prospective Randomized Phase II Study Assess the Schema of Retreatment With Lutathera® ([177LU]LU-DOTA-TATE) in Patients With New Progression of Intestinal Well-differenciated Neuroendocrine Tumor
Brief Title: Assessment of Retreatment With Lutathera® in Patients With New Progression of Intestinal Well-differenciated NET
Acronym: ReLUTH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2021-04 REL
Record Dates: First submitted 2021-06-11; First posted 2021-07-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors; Intestinal Well Differentiated Endocrine Tumor; Progressive Disease
MeSH Terms: conditions — Neuroendocrine Tumors; Disease Progression | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: It's a prospective, national, multicenter, open-label, randomized, phase II study, to compare 2 additional cycles of Lutathera® versus active surveillance in patients who already received two cycles of "Second PRRT" (already retreated with two cycles).
  Written informed consent will be collected before any study related procedures take place.
  Patients previously treated with 4 cycles of Lutathera® will be registered after a first progression (clinic, biologic and/or radiologic) of their neuroendocrine tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): 2 additional infusions of Lutathera® according to the marketing authorization schema
  Interventions: Drug: Lutathera
- Control arm (No Intervention): No treatment with active monitoring (clinical, biological and radiological follow-up) every 2 months.

INTERVENTIONS:
Drug: Lutathera — 2 additional infusions of Lutathera®
  Arms: Experimental arm

SUMMARY:
In France, since the reimbursement of Lutathera®, this treatment is allowed for retreatment if patients still fulfill the criteria of its indication and 4 news cycles could be proposed. However, clinical practices are heterogeneous regarding the number of new cycles and most teams perform only two additional cycles (every 8 weeks). Therefore, the coordinator propose to evaluate the efficacy of two additional cycle of Lutathera® versus active surveillance in patients already retreated with two cycles Lutathera® for a new progression of intestinal neuroendocrine tumor and who previously received the 4 cycles of treatment with a clinical benefit.

DETAILED DESCRIPTION:
The NETTER-1 clinical trial compared peptide receptor radionuclide therapy (PRRT) with [177Lu]Lu-DOTA-TATE (Lutathera®) every eight weeks (4 doses) plus 30 mg octreotide LAR every 4 weeks with high dose (60 mg) of octreotide LAR every 4 weeks in patients with progressive and unresectable midgut neuroendocrine well differentiated (G1, G2) tumors (NETs) with somatostatin-receptor positive imaging (SSTRi+). Lutathera® improves both median progression free survival (PFS) (28.4 months vs 8.5 months) and median overall survival (OS) ("not reached" vs 27.4 months) with a follow-up of 42 months. Lutathera® also has an impact on quality of life. Therefore, this treatment was approved by the European Medicines Agency and is now reimbursed in France in that specific indication. Despite these promising results, progression will occur in most of patients within a variable time with limited treatment options left. Retreatment with additional cycles of Lutathera® may be an option. Van der Zwan et al. showed in a large retrospective cohort (the "ROTTERDAM cohort") a median PFS of 14.6 months after retreatment with two additional cycles of PRRT with [177Lu]Lu-DOTA-TATE and a significant longer OS than in the non-randomized control group. Interestingly, the safety was similar in salvage group than in initial PRRT: no grade (G) 3/4 renal toxicity occurred and hematological toxicities were similar to the group of patients who received the initial treatment (4 cycles). In a smaller cohort of 15 patients, Yordanova et al. showed that 8 or more cycles of [177Lu]Lu-DOTA-TATE were well tolerated and led to a survival improvement. In this study, each salvage therapy consisted of 2 or 3 cycles. No severe (G3, G4) renal toxicity or G4 adverse event occurred. In France, since the reimbursement of Lutathera®, this treatment is allowed for retreatment if patients still fulfill the criteria of its indication and 4 news cycles could be proposed. However, clinical practices are heterogeneous regarding the number of new cycles and most teams perform only two additional cycles (every 8 weeks). Therefore, the coordinator propose to evaluate the efficacy of two additional cycle of Lutathera® versus active surveillance in patients already retreated with two cycles Lutathera® for a new progression of intestinal neuroendocrine tumor and who previously received the 4 cycles of treatment with a clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Histologically proven intestinal G1 or G2 neuroendocrine tumors (NET),
* Patient previously treated with 4 cycles of Lutathera® (defined as "First PRRT"),
* Disease control after "First PRRT" ≥ 12 months,
* Patient presenting a progression of disease (clinic, biologic and/or radiologic) after a first PRRT,
* Decision of retreatment with Lutathera® (defined as "Second PRRT") validated by RENATEN and/or multidisciplinary tumor board and in the scope of the French reimbursement process,
* ECOG performance status 0-2,
* Life expectancy ≥ 6 months as prognosticated by the physician,
* Somatostatin receptor imaging positive imaging (SSTRi+) disease within 4 months prior to inclusion : (may be PET imaging (68Ga-based SSTR analogues) or scintigraphy imaging: 111In-pentetreotide or 99mTc-octreotide. At least 90% of lesions must be positive for SSTRi with a significant uptake (>= liver of surrounding tissue),
* Measurable disease per RECIST 1.1 (Appendix 1), on CT/MRI scans, defined as at least 1 lesion with ≥ 1 cm in longest diameter, and ≥ 2 radiological tumors lesions in total,
* Adequate bone marrow reserve (Hb > 8 g/dl, neutrophils ≥ 1500/mm³ and platelets ≥ 80 000/mm³),
* Negative pregnancy test in women of childbearing potential (the β-HCG dosage must be ≤ 4 days before inclusion). Women who have no reproductive potential are postmenopausal women or women who have had permanent sterilization, eg. tubal occlusion, hysterectomy, bilateral salpingectomy),
* Effective contraception in men or women of childbearing or pre-menopausal age and up to a minimum of 6 months following the end of treatment,
* Patient´s signed written informed consent,
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures,
* Affiliation to the French Social Security System

Exclusion Criteria:

* Patient who did not respond (no CR, PR or SD) to "first PRRT".
* Radiological progression after two cycles of "Second PRRT" according to RECIST version 1.1,
* Grade 4 hematotoxicity and/or nephrotoxicity during the initial PRRT, or unresolved AEs categorized as Grade 2 or higher (as per Common Terminology Criteria for Adverse Events (CTCAE v5.0) from previous PRRT cycles or any other therapy for NET, excluding alopecia and peripheral neuropathy,
* Pancreatic NET,
* NeuroEndocrine Carcinoma,
* Prior external beam radiation therapy to more than 25% of the bone marrow,
* Severe renal (estimated Glomerular Filtration Rate (GFR) according to Modification of Diet in Renal Disease (MDRD) < 40 mL/min or nephrotic syndrome) or hepatic insufficiency (Alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) > 2.5 x ULN or ALT/AST > 5 x ULN if liver function abnormalities are due to the underlying malignancy and/or total serum bilirubin > 2.5 x ULN),
* Serum albumin < 3.0 g/dL unless prothrombin time is within the normal range,
* Uncontrolled diabetes mellitus as defined by a fasting blood glucose above 2 ULN,
* Uncontrolled decompensated heart failure, myocardial infarction uncontrolled, stroke, pulmonary embolism or revascularization procedure, unstable angina pectoris, uncontrolled cardiac arrhythmia, and clinically significant bradycardia during the last 12 months,
* Hypertension that cannot be controlled despite medications (≥ 160/95 mmHg despite optimal medical therapy)
* Brain metastases (unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrolment in the study. Patients with a history of brain metastases must have a head CT scan with contrast or MRI to document stable disease prior to enrolment in the study),
* Pregnancy or breast feeding,
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results,
* Known hypersensitivity to any of the study drugs, study drug classes, or any constituent of the products,
* Concomitant participation or participation within the last 30 days in another clinical trial,
* History of other solid tumor in 5 years before the inclusion excepted of cancer in situ of the cervix and skin cancer (basal or squamous cell) treated and controlled.
* Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of two additional cycles of Lutathera® (one injection every two months), compared to active surveillance during 6 months in patients already retreated with two cycles. | assessement every cycle (every 8 weeks) 6 months from randomization
  defined as a change of tumoral assessment (Complete Response, Partial Response and Stable Disease from RECIST v1.1) with an evaluation every 2 months.

SECONDARY OUTCOMES:
Evaluate the impact of two additional cycles of Lutathera® (one injection every two months), compared to active surveillance in term of Safety | during 6 months in patients already retreated with two cycles (each cycle is 8 weeks)
  Number and type of adverse event according to NCI-CTCAE v5.0.
Evaluate the impact of two additional cycles of Lutathera® (one injection every two months), compared to active surveillance in term of Progression free survival | the time without progression of disease during 5 years after the treatment,
  the time from randomization until documented disease progression on radiological tumor assessment (as evaluated by an independent central review by radiologists blindly of the treatment assignments according to RECIST v1.1) or death from any cause, whichever occurs first
Evaluate the impact of two additional cycles of Lutathera® (one injection every two months), compared to active surveillance in term of Overall survival | the time without death during 5 years after the treatment
  the time from randomization until death from any cause.
To assess quality of life of general patient | during and after treatment in both arm : every 8 wweks during the treatment, every 3 months during 1 year post treatment and every year during 4 years post treatment
  Quality of life will be measured by EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer, Quality-of-life questionnaire C30, no min and max values)
To assess quality of life of gastrointestinal neuroendocrine tumor | during and after treatment in both arm : every 8 wweks during the treatment, every 3 months during 1 year post treatment and every year during 4 years post treatment
  Quality of life will be measured by EORTC GI.NET21 questionnaire (European Organisation for Research and Treatment of Cancer, gastrointestinal neuroendocrine tumor, no min and max values)

CONTACTS AND LOCATIONS:
Overall Officials: Deshayes Emmanuel, PHD, Study Chair — ICM Co. Ltd.
Locations (28):
- France (28):
  - Institut de Cancérologie de l'Ouest Site d'Angers, Angers
  - Institut Bergonié, Bordeaux
  - CHRU Morvan, Brest
  - Hospices civils de LYON - GHE, Bron
  - Centre François Baclesse, Caen
  - CH Métropole de Savoie, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - CHU de DIJON, Dijon
  - CHU Grenoble Alpes (CHUGA), La Tronche
  - CHRU Lille, Lille
  - Centre léon bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de la Timone, Marseille
  - ICM Val d'Aurelle, Montpellier
  - CHU Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Pitié Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Henri Becquerel, Rouen
  - CHU de Rouen, Rouen
  - CHU ST Etienne, Saint-Etienne
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de cancérologie Strasbourg, Strasbourg
  - IUCT Oncopole, Toulouse
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after coding by an inclusion number, 1st letter of the surname and first name can be shared.
  Participant data will be available upon request and with the completion of a contract between the sponsor and the applicant.
  The study protocol, the statistical analysis plan and the analytical code may also be subject to data sharing under a transfer contract (EU-MCR).

REFERENCES:
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Strosberg J, El-Haddad G, Wolin E, Hendifar A, Yao J, Chasen B, Mittra E, Kunz PL, Kulke MH, Jacene H, Bushnell D, O'Dorisio TM, Baum RP, Kulkarni HR, Caplin M, Lebtahi R, Hobday T, Delpassand E, Van Cutsem E, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Oberg K, Lopera Sierra M, Santoro P, Thevenet T, Erion JL, Ruszniewski P, Kwekkeboom D, Krenning E; NETTER-1 Trial Investigators. Phase 3 Trial of 177Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med. 2017 Jan 12;376(2):125-135. doi: 10.1056/NEJMoa1607427. PMID 28076709
- [Background] Strosberg J, Wolin E, Chasen B, Kulke M, Bushnell D, Caplin M, Baum RP, Kunz P, Hobday T, Hendifar A, Oberg K, Sierra ML, Thevenet T, Margalet I, Ruszniewski P, Krenning E; NETTER-1 Study Group. Health-Related Quality of Life in Patients With Progressive Midgut Neuroendocrine Tumors Treated With 177Lu-Dotatate in the Phase III NETTER-1 Trial. J Clin Oncol. 2018 Sep 1;36(25):2578-2584. doi: 10.1200/JCO.2018.78.5865. Epub 2018 Jun 7. PMID 29878866
- [Background] Rudisile S, Gosewisch A, Wenter V, Unterrainer M, Boning G, Gildehaus FJ, Fendler WP, Auernhammer CJ, Spitzweg C, Bartenstein P, Todica A, Ilhan H. Salvage PRRT with 177Lu-DOTA-octreotate in extensively pretreated patients with metastatic neuroendocrine tumor (NET): dosimetry, toxicity, efficacy, and survival. BMC Cancer. 2019 Aug 8;19(1):788. doi: 10.1186/s12885-019-6000-y. PMID 31395036
- [Background] Vaughan E, Machta J, Walker M, Toumpanakis C, Caplin M, Navalkissoor S. Retreatment with peptide receptor radionuclide therapy in patients with progressing neuroendocrine tumours: efficacy and prognostic factors for response. Br J Radiol. 2018 Nov;91(1091):20180041. doi: 10.1259/bjr.20180041. Epub 2018 Mar 20. PMID 29513039
- [Background] Yordanova A, Mayer K, Brossart P, Gonzalez-Carmona MA, Strassburg CP, Essler M, Ahmadzadehfar H. Safety of multiple repeated cycles of 177Lu-octreotate in patients with recurrent neuroendocrine tumour. Eur J Nucl Med Mol Imaging. 2017 Jul;44(7):1207-1214. doi: 10.1007/s00259-017-3652-1. Epub 2017 Mar 1. PMID 28246882
- [Background] Sabet A, Haslerud T, Pape UF, Sabet A, Ahmadzadehfar H, Grunwald F, Guhlke S, Biersack HJ, Ezziddin S. Outcome and toxicity of salvage therapy with 177Lu-octreotate in patients with metastatic gastroenteropancreatic neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2014 Feb;41(2):205-10. doi: 10.1007/s00259-013-2547-z. Epub 2013 Sep 13. PMID 24030668
- [Background] van Essen M, Krenning EP, Kam BL, de Herder WW, Feelders RA, Kwekkeboom DJ. Salvage therapy with (177)Lu-octreotate in patients with bronchial and gastroenteropancreatic neuroendocrine tumors. J Nucl Med. 2010 Mar;51(3):383-90. doi: 10.2967/jnumed.109.068957. Epub 2010 Feb 11. PMID 20150247
- [Background] Gleisner KS, Brolin G, Sundlov A, Mjekiqi E, Ostlund K, Tennvall J, Larsson E. Long-Term Retention of 177Lu/177mLu-DOTATATE in Patients Investigated by gamma-Spectrometry and gamma-Camera Imaging. J Nucl Med. 2015 Jul;56(7):976-84. doi: 10.2967/jnumed.115.155390. Epub 2015 May 21. PMID 25999429
- [Background] Sundlov A, Sjogreen-Gleisner K, Svensson J, Ljungberg M, Olsson T, Bernhardt P, Tennvall J. Individualised 177Lu-DOTATATE treatment of neuroendocrine tumours based on kidney dosimetry. Eur J Nucl Med Mol Imaging. 2017 Aug;44(9):1480-1489. doi: 10.1007/s00259-017-3678-4. Epub 2017 Mar 22. PMID 28331954
- [Background] Del Prete M, Buteau FA, Arsenault F, Saighi N, Bouchard LO, Beaulieu A, Beauregard JM. Personalized 177Lu-octreotate peptide receptor radionuclide therapy of neuroendocrine tumours: initial results from the P-PRRT trial. Eur J Nucl Med Mol Imaging. 2019 Mar;46(3):728-742. doi: 10.1007/s00259-018-4209-7. Epub 2018 Nov 30. PMID 30506283
- [Background] Deshayes E, Assenat E, Meignant L, Bardies M, Santoro L, Gourgou S. A prospective, randomized, phase II study to assess the schemas of retreatment with Lutathera(R) in patients with new progression of an intestinal, well-differentiated neuroendocrine tumor (ReLUTH). BMC Cancer. 2022 Dec 22;22(1):1346. doi: 10.1186/s12885-022-10443-4. PMID 36550428
- See also: RCP — https://www.ema.europa.eu/en/documents/product-information/lutathera-epar-product-information_fr.pdf
- See also: HAS — https://www.has-sante.fr/jcms/pprd_2983166/fr/lutathera-lutecium-177lu-oxodotreotide